CLINICAL TRIAL: NCT06318897
Title: Open-label, Single Center, Single-arm, Phase 2 Study of Neoadjuvant Pembrolizumab in Combination With Carboplatin and Paclitaxel in Patients With Stage 1 cT1b-T1cN0M0 Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0645; NCI-2024-02384 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Stage 1 cT1b-T1cN0M0; Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; pembrolizumab; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pathologic Complete Response (Experimental): If a participant's tissue shows a pathological complete response to treatment, participants will receive up to 13 cycles of pembrolizumab alone. Pathological complete response means that the study team cannot find any evidence of cancer in the breast or lymph node tissue sample that was removed during the participants surgery, after the participant completes the 4 cycles of carboplatin, pembrolizumab and paclitaxel.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pembrolizumab
- Non-Pathologic Complete Response (Experimental): If a participant's tissue does not show a pathological complete response, the participant will receive 4 cycles of pembrolizumab plus 2 other drugs (doxorubicin and cyclophosphamide), followed by 9 cycles of pembrolizumab alone.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pembrolizumab; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Carboplatin — Given by IV
  Other Names: Paraplatin®
Drug: Paclitaxel — Given by IV
  Other Names: PACLITAXEL PROTEIN BOUND
Drug: Pembrolizumab — Given by IV
  Other Names: KEYTRUDA®
Drug: Doxorubicin — Given by IV
  Other Names: Doxorubicin Hydrochloride; Adriamycin PFS®; Adriamycin RDF™; Adriamycin®; Rubex®
  Arms: Non-Pathologic Complete Response
Drug: Cyclophosphamide — Given by IV
  Other Names: Cytoxan®; Neosar®
  Arms: Non-Pathologic Complete Response

SUMMARY:
To look at the effectiveness of the combination of pembrolizumab, carboplatin, and paclitaxel in participants with stage 1 cT1b-T1cN0M0 Triple Negative Breast Cancer.

DETAILED DESCRIPTION:
Primary Objective To estimate the rate of pCR in patients with cT1b and T1cN0M0 TNBC after neoadjuvant therapy with 4 cycles of Pembrolizumab + Carboplatin + Paclitaxel.

Secondary Objective To assess the safety and toxicity profile of pembrolizumab plus chemotherapy in participants receiving an anthracycline-de-escalated regimen of carboplatin, paclitaxel and pembrolizumab by recording the incidence of treatment emergent adverse events.

Exploratory Objectives

1. To estimate the invasive disease-free survival (iDFS), and overall survival (OS) in participants with cT1b-T1cN0 TNBC that receive neoadjuvant pembrolizumab plus chemotherapy in the setting of an anthracycline de-escalation study.
2. To explore if there is a molecular signature associated with response or lack of response to therapy.
3. To evaluate patient reported outcomes of participants receiving this de-escalated regimen.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participants must have histologically confirmed ER negative, PR negative and HER2-negative (TNBC) defined as ER<10%, PR<10%, and HER2 negative (per 2018 ASCO CAP guidelines). All pathology will be confirmed at the MD Anderson Houston Campus. Participants with tumors designated as HER2 equivocal (per ASCO CAP guidelines) are eligible if in view of treating physician patient is not considered a candidate for HER2-targeted therapy. Participants with weakly ER or PR positive disease, defined as ER and/or PR between 1-9% by immunohistochemistry, are eligible if the treating physician considers the participants not eligible for adjuvant endocrine therapy.
2. AJCC 8 anatomic tumor Stage 1 T1b-T1c, N0, M0. All participants with clinically suspicious nodes must undergo core or fine needle biopsy per standard clinical practice to pathologically assess at least 1 suspicious index node. Participants with suspicious nodes that are biopsy negative will be eligible.
3. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of Stage 1 T1b-T1cN0M0 TNBC will be enrolled in this study.
4. Male participants: A male participant must agree to use a contraception as detailed in Appendix 2 of this protocol during the treatment period and for at least 120 days, corresponding to time needed to eliminate any study treatment(s) (e.g. 5 terminal half-lives for pembrolizumab and/or any active comparator/combination) plus an additional 90 days (a spermatogenesis cycle) for study treatments with evidence of genotoxicity at any dose after the last dose of study treatment and refrain from donating sperm during this period.
5. Female participants: A female participant is eligible to participate if she is not pregnant (see Appendix 2), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 2 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 2 during the treatment period and for at least 120 days (corresponding to time needed to eliminate any study treatment(s) (pembrolizumab and/or any active comparator/combination) plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity after the last dose of study treatment.
6. Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible.
7. The participant provides written informed consent for the trial.
8. Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 (appendix 3). Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
10. Have adequate organ function as defined in the following table (Table 3). Specimens must be collected within 10 days prior to the start of study intervention.
11. Non-English speaking participant can enroll in the study as long as they speak a language for which interpretation can be provided by a licensed interpreter either in person or virtually.
12. Criteria for known HIV positive participants.

    1. Participants with HIV are eligible if they have well-controlled HIV with negative viral load on ART and must not have had any AIDS-defining opportunistic infections within the past 12 months from initiation of C1D1 study treatment.
    2. HIV screening tests are not required unless:

    i. Known history of HIV ii. As mandated by local health authority
13. Criteria for known Hepatitis B and C positive participants Hepatitis B and C screening tests are not required unless:

    * Known history of HBV or HCV infection
    * As mandated by local health authority 13.1 Hepatitis B positive Participants
    * Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.
    * Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention. 13.2 Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.
    * Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

Table 3 Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) = ≥1500/µL Platelets = ≥100 000/µL Hemoglobin = ≥9.0 g/dL or ≥5.6 mmol/La Renal Creatinine OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) = ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN Hepatic Total bilirubin = ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT) = ≤2.5 × ULN (≤5 × ULN for participants with liver metastases) Coagulation International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) = ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal. a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks. b Creatinine clearance (CrCl) should be calculated per institutional standard. Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Stage 2, 3 or 4 Triple negative breast cancer
2. Hormone Receptor positive and/or Human Epidermal Growth factor 2 (HER 2) positive breast cancer
3. A WOCBP who has a positive urine pregnancy test within 72 hours prior to dose of study drug (see Appendix 2). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
5. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks to allocation of therapy.
6. Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease, with a 1-week washout, is permitted.
7. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
8. Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
11. Has known active CNS metastases and/or carcinomatous meningitis.
12. Has severe hypersensitivity (≥Grade 3) to any of the components or any of its excipients used in the study treatments.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
14. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
15. Has an active infection requiring systemic therapy for >14 days from initiation of C1D1 study treatment.
16. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection. Note: Hepatitis B and C screening tests are not required unless:

    * Known history of HBV and HCV infection
    * As mandated by local health authority
17. Has not adequately recovered from major surgery or has ongoing surgical complications.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
21. Has had an allogenic tissue/solid organ transplant.
22. Participants with the following contraindications to doxorubicin therapy: recent myocardial infarction; severe myocardial insufficiency; severe arrhythmias; previous treatment with complete cumulative doses of doxorubicin, daunorubicin, idarubicin, and/or other anthracyclines and anthracenedione.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Oluchi Oke, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org